CLINICAL TRIAL: NCT01555918
Title: A Phase I, Open-Label, Single and Multiple Dose Study to Assess the Safety and Pharmacokinetics of Isavuconazole in Healthy Chinese Volunteers
Brief Title: A Study to Assess the Safety and Pharmacokinetics of Isavuconazole in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 9766-CL-0038
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Pharmacokinetics of BAL4815; Pharmacokinetics of BAL8728; Healthy Volunteers
Keywords: Pharmacokinetics; Healthy volunteers; Isavuconazole; BAL4815; BAL8728; BAL8557
MeSH Terms: interventions — isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Isavuconazole single oral dose - Part 1 (Experimental)
  Interventions: Drug: Isavuconazole
- Isavuconazole single intravenous (IV) dose - Part 1 (Experimental)
  Interventions: Drug: Isavuconazole (IV)
- Isavuconazole multiple oral doses - Part 2 (Experimental)
  Interventions: Drug: Isavuconazole
- Isavuconazole multiple intravenous (IV) doses -Part 2 (Experimental)
  Interventions: Drug: Isavuconazole (IV)

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: BAL4815, BAL8557, BAL8728
  Arms: Isavuconazole multiple oral doses - Part 2; Isavuconazole single oral dose - Part 1
Drug: Isavuconazole (IV) — intravenous (IV)
  Other Names: BAL4815, BAL8557, BAL8728
  Arms: Isavuconazole multiple intravenous (IV) doses -Part 2; Isavuconazole single intravenous (IV) dose - Part 1

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic properties of isavuconazole (BAL4815) and the cleavage product (BAL8728) and assess the safety and tolerability after single-dose and steady state (multiple-dose) administration of isavuconazole BAL8557 in healthy Chinese subjects.

DETAILED DESCRIPTION:
This is a two part study:

Part 1: On Day 1, Period 1, subjects will receive a single dose of isavuconazole orally or intravenously according to the treatment sequence allocation. Subjects will remain resident in the unit in order to collect blood for pharmacokinetics (PK) and to assess the safety tests. They will be released in the morning of Day 15 after collection of blood for safety tests. Subjects will have a washout period of 2 weeks returning to the unit for Day -1 of Period 2 (Day 29). Subjects will receive a single dose of isavuconazole orally or intravenously (opposite mode of administration from Period 1). Subjects will remain resident in the unit and will be released in the morning of Day 15, Period 2 (Day 44) after collection of blood for tests.

Part 2: Subjects will be allocated to multiple intravenous (IV) (Group 1) or oral (Group 2) dosing. On Day 1, Group 1 will receive multiple intravenous (IV) dosing of isavuconazole as a 2-hour infusion, three times a day (TID) with 8 hours between doses for 2 days followed by isavuconazole as a 2-hour infusion every day (QD) for 10 days. Group 2 will receive multiple oral (PO) dosing of isavuconazole TID with 8 hours between doses for 2 days followed by isavuconazole PO QD for 10 days. Subjects in Group 1 and 2 will remain resident in the unit in order to collect blood and urine for PK evaluations and to assess the safety tests. They will be released in the morning of Day 26 after collection of blood for tests.

ELIGIBILITY:
Inclusion Criteria:

* The subject weighs at least 50 kg, and has a body mass index of 19 to 24 kg/m2 inclusive.
* The subject's 12-lead electrocardiogram (ECG) is normal
* The subject's physical examination and clinical laboratory test results are within normal limits
* If female, the subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years without menses), or using a medically acceptable double-barrier method (e.g. spermicide and diaphragm, spermicide and condom) to prevent pregnancy and agrees to continue using this method from Screening until the end of study; and is not lactating or pregnant as documented by negative serum pregnancy tests
* If male, the subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy during the study period.
* The subject agrees to comply with diet and smoking restrictions prior to entry in the clinical unit, during confinement and until the end of the study.
* The subject has good venous access.

Exclusion Criteria:

* The subject has a history of any clinically significant cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy with the exception of non-melanoma skin cancer.
* The subject has a history of gastrointestinal tract surgery.
* The subject has a known or suspected hypersensitivity to isavuconazole, the azole class of compounds or any components of the study drug.
* The subject has a history of consuming more than 14 units of alcoholic beverages per week, has a history of drug or alcohol abuse within the past 2 years or has a positive screen for alcohol or drugs of abuse/illegal drugs (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits).
* The subject uses tobacco containing products or nicotine containing products of more than 5 cigarettes/day or the equivalent amount of tobacco.
* The subject is positive for human immunodeficiency virus antibody or Treponema pallidum.
* The subject is positive for hepatitis C antibody or hepatitis B antigen
* The subject consumes more than 1 liter of tea and coffee per day and anticipates an inability to abstain from caffeine or alcohol use for 48 hours prior to clinic admission on Day -1 and throughout the duration of the study; or from grapefruit, Seville oranges, star fruit, or any products containing these items from 72 hours prior to clinic admission on Day -1 and throughout the duration of the study.
* The subject has been vaccinated within 30 days or has had treatment with prescription drugs or over-the-counter medications (including complementary and alternative medicines) within 14 days prior to Check-in (Day -1), with the exception of paracetamol up to 2g/day but not more than 4 days/week (depot preparations are prohibited).
* The subject has participated in other clinical trials within 2 months prior to study drug administration.
* The subject has donated or had any significant blood loss over 200 mL, or received a transfusion of any blood or blood products within 2 months prior to Day 1.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetics of isavuconazole in plasma (Part 1): Cmax, AUClast, AUCinf, AUC24, tmax, t1/2, CL/F, Vz/F, F, MRT, CLtot, and Vz | Day 1 to Day 15 in each treatment period (19 time points)
  Cmax, AUC from the time of dosing to the last quantifiable concentration (AUClast), AUC from time 0 extrapolated to infinity (AUCinf), AUC from time 0 to 24 hours (AUC24), Time to attain Cmax (tmax), Apparent Terminal Elimination Half-Life (t1/2), Apparent body clearance after extravascular dosing (CL/F), Apparent volume of distribution during the terminal phase after single or repeated extravascular dosing (Vz/F), Bioavailability (F), Mean residence time (MRT), Total body clearance after intravenous (IV) dosing (CLtot), Volume of distribution during the terminal phase after IV dosing (Vz)
Composite of pharmacokinetics of isavuconazole in plasma (Part 2): Cmax, Cmin, AUCtau, tmax, t1/2, CL/F, Vz/F, PTR, CLtot, MRT, and Vss | Day 1 to Day 26 (33 time points)
  Cmax, Minimum observed concentration (Cmin), AUC during the time interval between consecutive dosing (AUCtau), Time to attain Cmax (tmax), Apparent Terminal Elimination Half-Life (t1/2), Apparent body clearance after extravascular dosing (CL/F), Apparent volume of distribution during the terminal phase after single or repeated extravascular dosing (Vz/F), Peak trough fluctuation within one dosing interval at steady state (PTR), Total body clearance after intravenous (IV) dosing (CLtot), Mean residence time (MRT), Volume of distribution at steady state determined after IV dosing (Vss)
Composite of pharmacokinetics of isavuconazole in urine (Part 2): Cumulative amount of drug excreted over the time interval between consecutive dosing (Aetau), Fraction of Aetau (Aetau %), Renal clearance (CLR) | Day 12 (2 time points)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Huashan Hospital, Shanghai, China